CLINICAL TRIAL: NCT03474016
Title: The Role of Circulating Cell-free DNA and Its Integrity Using ALU (247/115) bp Sequences as a Biomarker for Diagnosis of Breast Cancer
Brief Title: Cell Free DNA and Its Integrity Using ALU Sequences as a Biomarker for Diagnosis of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Mostafa Mohamed, Principle investigator, Assiut University
Other Study IDs: CFDAIIUASABFDOBC
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with early breast cancer(30)
  Interventions: Diagnostic Test: Mammography-Histopathological examination of breast mass specimens- polymerase chain reaction
- Patients with advanced breast cancer(30)
  Interventions: Diagnostic Test: Mammography-Histopathological examination of breast mass specimens- polymerase chain reaction
- Patients with benign breast diseases(20)
  Interventions: Diagnostic Test: Mammography-Histopathological examination of breast mass specimens- polymerase chain reaction
- Apparently healthy females as a control group(36)
  Interventions: Diagnostic Test: Mammography-Histopathological examination of breast mass specimens- polymerase chain reaction

INTERVENTIONS:
Diagnostic Test: Mammography-Histopathological examination of breast mass specimens- polymerase chain reaction — Mammography-Histopathological examination of breast mass specimens-Detection of long and short DNA fragments in serum using real-time quantitative polymerase chain reaction

SUMMARY:
Breast cancer (BC) is the most common cancer in women worldwide, and is the leading cause of death from cancer among women globally. Mammography is the standard method for early detection of BC in many countries, with over 1.3 million annually new diagnosed cases.In Egypt, breast cancer is the most common cancer in females accounting for 38.8% of all female cancers.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common cancer in women worldwide, and is the leading cause of death from cancer among women globally. Mammography is the standard method for early detection of BC in many countries, with over 1.3 million annually new diagnosed cases.In Egypt, breast cancer is the most common cancer in females accounting for 38.8% of all female cancers. Whereas radiological screening programs have been successfully applied in detecting breast cancer in earlier stages, no valuable blood biomarkers have been yet identified for that purpose. However, false-positive recall rates vary according to age, breast density, and postmenopausal hormonal therapy, among other. For women with dense breasts, the accuracy of mammography is decreased. Circulating serum marker for monitoring of BC have been in development for several decades. Conventional tumor markers, such as cancer antigen 15-3 (CA15-3), carcinoembryonic antigen (CEA)), and circulating tumor cell count (CTC), are clinically available, however, their usefulness is mostly limited to patients with advanced and metastatic BC (MBC). Hence, there is a need for developing new biomarkers which can be used as valuable tools in identifying high risk patients, to predict disease prognosis and thus have an impact in patient management.Cell free DNA (cfDNA) are short fragments of nucleic acids present in the circulation. Multiple studies also have indicated elevated levels of cf DNA in breast cancer. The ALU(Arthrobacter luteus) sequences were chosen, as they are the most abundant and active repeated elements in the human genome, typically 300 nucleotides in length, accounting for more than 10% of the genome. DNA integrity was calculated as the ratio of (ALU247/ALU115). As the annealing sites of ALU115 are within the ALU247 annealing sites, thus the ratio of ALU247 to ALU115 is termed as DNA integrity. It characterizes the fragmentation pattern of circulating cell free DNA. The DNA integrity is "1" if template DNA is not truncated and "0" if DNA is completely truncated to fragments smaller than 247 bp (base pair). Thus it has been assessed for its diagnostic and prognostic potential role in breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled before initiation of any treatment.

Exclusion Criteria:

* Any other malignant or benign tumors.
* Active inflammatory or autoimmune diseases.
* Renal or liver diseases.

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study will be conducted on one hundred informed and consented female individuals (according to the guidelines of ethical committee of faculty of Medicine, Assuit University and South Egypt Cancer Institute.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic values of cell free DNA using ALU (Arthrobacter luteus) sequence levels (247 bp (base pair), 115bp) and its integrity in peripheral blood of breast cancer patients as non invasive marker. | 3 days